CLINICAL TRIAL: NCT03044743
Title: A Phase I/II Trial of PD-1 Knockout EBV-CTLs for Advanced Stage EBV Associated Malignancies
Brief Title: PD-1 Knockout EBV-CTLs for Advanced Stage Epstein-Barr Virus (EBV) Associated Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yang Yang (Other)
Responsible Party: Sponsor-Investigator, Yang Yang, MD, PhD, MSCR, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-1-KO-EBV-CTL
Record Dates: First submitted 2017-01-22; First posted 2017-02-07 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Stage IV Gastric Carcinoma; Stage IV Nasopharyngeal Carcinoma; T-Cell Lymphoma Stage IV; Stage IV Adult Hodgkin Lymphoma; Stage IV Diffuse Large B-Cell Lymphoma
Keywords: PD-1; CRISPR Cas9; EBV; advanced stage malignancies
MeSH Terms: conditions — Stomach Neoplasms; Nasopharyngeal Carcinoma; Lymphoma, T-Cell; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 knockout EBV-CTL (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISP-Cas9 system and EBV-CTL will be generated in the laboratory (PD-1 Knockout EBV-CTL).
  Fludarabine at 30mg/m2 and Cyclophosphamide at 300mg/m2 single dose will be administered 3 days i.v. before cell infusion.
  A total of 2 x 10^7/kg PD-1 Knockout CTL will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third.
  Interleukin-2 (IL-2) will be given daily( iv) since the first day of the cell infusion for 5 consecutive days, 4000,000 international unit（IU）/day . Patients will receive a total of four cycles of treatment.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Interleukin-2

INTERVENTIONS:
Drug: Fludarabine — To modify immune micro-environment
  Other Names: Fludara
Drug: Cyclophosphamide — To modify immune micro-environment
  Other Names: Cytoxan
Drug: Interleukin-2 — To sustain the survival of infused T cells
  Other Names: IL-2

SUMMARY:
This study will evaluate the safety of PD-1 knockout EBV-CTL cells in treating EBV (Epstein-Barr virus) positive advanced stage malignancies. Blood samples will also be collected for research purposes.

DETAILED DESCRIPTION:
This is a study of CRISPR-Cas9 mediated PD-1 knockout-T cells from autologous origin. Patients are assigned to receive 4 circles of cell therapy. The safety and clinical response are evaluated. Biomarkers and immunological markers are also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically verified stage IV gastric carcinoma, nasopharyngeal carcinoma and lymphoma with measurable lesions (At least one measurable lesion or the immunotherapy)
* Pathologically verified as EBV positive malignancies
* Human leukocyte antigen (HLA) genotypes: HLA-A02, HLA-A24 or HLA-A11 genotypes
* Progressed after standard treatment or the patients refused to accept the standard treatment
* Performance score: 0-1
* Expected life span: >= 3 months
* Toxicities from prior treatment has resolved. Washout period is 1 months
* Major organs function normally
* Women at pregnant ages should be under contraception
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients with possible drug allergy of immunotherapy
* Patients with active bacterial or fungal infections
* Coagulopathy, or ongoing thrombolytics and/or anticoagulation
* Blood-borne infectious disease, e.g. hepatitis B, hepatitis C and HIV
* History of coronary artery disease, asthma, or vascular disease or other disease inappropriate for treatment deemed by treating physician
* With other tumors except for in situ cervical cancer, treated squamous cell carcinoma and bladder cancer (Ta and TIS) or other malignancies that have been treated with radical therapy (at least for 5 years before the enrollment)
* With other immune diseases, or chronic use of immunosuppressants or steroids
* Pregnant and lactating women
* Compliance cannot be expected
* Other conditions requiring exclusion deemed by physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-04-07 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events using Common Terminology Criteria for Adverse Events (CTCAE v4.0) in patients | 6 months

SECONDARY OUTCOMES:
Response Rate | 90 days
Progression free survival (PFS) | up to 1 year
Overall Survival (OS) | up to 3 years
The duration of the normalization of tumor marker | up to 3 years
Interferon-γ change of T cells in the peripheral blood stimulated by tumor antigens | Baseline and 1 month, 3 months and 6 months
Th1/Th2 change in the peripheral blood | Baseline and 1 month, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Baorui Liu, MD, Principal Investigator — The Comprehensive Cancer Centre of Drum Tower Hospital, Medical School of Nanjing University and Clinical Cancer Institute of Nanjing University
Locations (1):
- The Comprehensive Cancer Center of Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim SY, Park C, Kim HJ, Park J, Hwang J, Kim JI, Choi MG, Kim S, Kim KM, Kang MS. Deregulation of immune response genes in patients with Epstein-Barr virus-associated gastric cancer and outcomes. Gastroenterology. 2015 Jan;148(1):137-147.e9. doi: 10.1053/j.gastro.2014.09.020. Epub 2014 Sep 22. PMID 25254613
- [Background] Quan L, Chen X, Liu A, Zhang Y, Guo X, Yan S, Liu Y. PD-1 Blockade Can Restore Functions of T-Cells in Epstein-Barr Virus-Positive Diffuse Large B-Cell Lymphoma In Vitro. PLoS One. 2015 Sep 11;10(9):e0136476. doi: 10.1371/journal.pone.0136476. eCollection 2015. PMID 26361042
- [Background] Louis CU, Straathof K, Bollard CM, Ennamuri S, Gerken C, Lopez TT, Huls MH, Sheehan A, Wu MF, Liu H, Gee A, Brenner MK, Rooney CM, Heslop HE, Gottschalk S. Adoptive transfer of EBV-specific T cells results in sustained clinical responses in patients with locoregional nasopharyngeal carcinoma. J Immunother. 2010 Nov-Dec;33(9):983-90. doi: 10.1097/CJI.0b013e3181f3cbf4. PMID 20948438
- [Background] Lloyd A, Vickery ON, Laugel B. Beyond the antigen receptor: editing the genome of T-cells for cancer adoptive cellular therapies. Front Immunol. 2013 Aug 5;4:221. doi: 10.3389/fimmu.2013.00221. eCollection 2013. PMID 23935598
- [Background] Su S, Hu B, Shao J, Shen B, Du J, Du Y, Zhou J, Yu L, Zhang L, Chen F, Sha H, Cheng L, Meng F, Zou Z, Huang X, Liu B. CRISPR-Cas9 mediated efficient PD-1 disruption on human primary T cells from cancer patients. Sci Rep. 2016 Jan 28;6:20070. doi: 10.1038/srep20070. PMID 26818188
- [Background] Mali P, Esvelt KM, Church GM. Cas9 as a versatile tool for engineering biology. Nat Methods. 2013 Oct;10(10):957-63. doi: 10.1038/nmeth.2649. PMID 24076990